CLINICAL TRIAL: NCT01656096
Title: Renal Sympathetic Denervation in Patients With Mild Refractory Hypertension
Brief Title: Renal Sympathetic Denervation in Mild Refractory Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Steffen Desch, MD, Principal Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSD-Leipzig
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Refractory Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal sympathetic denervation (Experimental): Renal sympathetic denervation (Symplicity ablation catheter, Medtronic Inc. Minneapolis, Minnesota, USA)
  Interventions: Device: Renal sympathetic denervation (Symplicity ablation catheter, Medtronic Inc. Minneapolis, Minnesota, USA)
- Sham procedure (Sham Comparator): Sham procedure mimicking the renal sympathetic denervation procedure in the experimental arm
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: Renal sympathetic denervation (Symplicity ablation catheter, Medtronic Inc. Minneapolis, Minnesota, USA)
  Arms: Renal sympathetic denervation
Other: Sham procedure
  Arms: Sham procedure

SUMMARY:
The purpose of this study is to examine the benefit of renal sympathetic denervation in patients with mild refractory hypertension

ELIGIBILITY:
Inclusion Criteria:

* Refractory hypertension: 3 or more antihypertensive agents of different classes (including a diuretic) at optimal dosage without change in the 4 weeks preceding randomization
* Systolic blood pressure of 135-149 and/or diastolic blood pressure of 90-94 mmHg (ABPM mean daytime values)
* No change in blood pressure medication within 6 months after randomization
* Age 18 to 75 years
* Informed consent

Exclusion Criteria:

* Blood pressure outside range mentioned above
* Renal, aortic or pelvic anatomy unsuited for renal sympathetic denervation
* Estimated glomerular filtration rate <45 mL/min/1.73 m² (modification of diet in renal disease formula)
* Unstable angina pectoris
* Myocardial infarction within 6 months prior to randomization
* Planned surgery or cardiovascular intervention within 6 months after randomization
* Severe heart valve disease
* Severe comorbidities with limited life expectancy
* Pregnancy
* Participation in another trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure (ABPM mean value) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Desch, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] Desch S, Okon T, Heinemann D, Kulle K, Rohnert K, Sonnabend M, Petzold M, Muller U, Schuler G, Eitel I, Thiele H, Lurz P. Randomized sham-controlled trial of renal sympathetic denervation in mild resistant hypertension. Hypertension. 2015 Jun;65(6):1202-8. doi: 10.1161/HYPERTENSIONAHA.115.05283. Epub 2015 Mar 30. PMID 25824248
- See also: Publication of study — http://www.ncbi.nlm.nih.gov/pubmed/25824248